CLINICAL TRIAL: NCT07377864
Title: Clinical Characteristics and Immune Escape Mechanism of Nontuberculous Mycobacterial Lung Disease in South China
Acronym: NTM-LD
Status: Not yet recruiting | Type: Observational
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-184-01
Record Dates: First submitted 2025-12-29; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Nontuberculous Mycobacterial Lung Disease; Mycobacterium Avium Complex (MAC)
Keywords: Nontuberculous Mycobacterial; South China; Immune Escape; Outcome
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMCs) and bronchoalveolar lavage fluid (BALF) cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective NTM Cohort: This cohort consists of approximately 1,500 patients diagnosed with nontuberculous mycobacterial (NTM) across multiple hospitals in South China. Data, including demographics, clinical symptoms, imaging findings, microbiology results, and treatment outcomes, will be extracted retrospectively from electronic medical records for the period from January 2015 to May 2025.
  Interventions: Other: Prospective Biospecimen Sub-cohort

INTERVENTIONS:
Other: Prospective Biospecimen Sub-cohort — Observational

SUMMARY:
Nontuberculous Mycobacterial lung disease (NTM-LD) is a significant infectious challenge. The precise causes remain unclear, diagnosis can be complex, treatment outcomes are often unsatisfactory, and the disease can severely affect a patient's quality of life. Environmental factors, such as the warm and humid climate in South China, may contribute to unique characteristics of NTM in this region, but systematic research is currently lacking.

This study aims to improve the understanding of NTM-LD in South China. It consists of two complementary parts:

1. The first part is a retrospective review of medical records from approximately 1,500 NTM patients across multiple hospitals in South China. This analysis seeks to identify common patterns in symptoms, diagnostic findings, and treatment responses within this population.
2. The second part is a prospective study involving about 106 current NTM-LD patients. Blood and lung fluid samples will be collected to analyze, using advanced laboratory techniques, how the patient's immune system responds to the infection. This investigation aims to uncover clues about why some cases are difficult to treat.

The overall goal of this research is to generate evidence that can aid healthcare providers in South China in diagnosing and managing NTM-LD more effectively. Please note that this is an observational study; no new drugs or experimental treatments are being tested.

DETAILED DESCRIPTION:
1. Background and Rationale NTM-LD presents significant clinical challenges due to its unclear pathogenesis, diagnostic complexity, suboptimal treatment outcomes, and poor prognosis. The unique climatic (hot, humid) and demographic factors in South China suggest potential regional variations in NTM epidemiology and clinical presentation. However, a systematic investigation into its clinical characteristics and underlying mechanisms in this region is lacking, impeding the development of localized precision medicine strategies.
2. Study Objectives Primary Objective: To systematically characterize the epidemiological patterns, clinical phenotypes, and prognostic determinants of NTM-LD in the South China population.

   Secondary Objectives:

   To analyze the distribution of NTM species and their correlation with disease severity and radiological findings.

   To investigate host immune microenvironment alterations post-NTM infection, focusing on inflammatory responses and immune cell functional states.

   To explore molecular mechanisms associated with treatment refractoriness in NTM disease.
3. Study Design

   This is a hybrid observational study comprising two distinct parts:
   * Part 1: A multicenter, retrospective, non-interventional survey study.
   * Part 2: A prospective observational study involving biospecimen collection and laboratory analysis.
4. Study Populations and Sample Size

   * Part 1: Approximately 1,500 patients diagnosed with NTM lung disease per standard guidelines between January 2015 and May 2025 across multiple collaborating centers in South China.
   * Part 2: A subset of 106 consecutively enrolled, confirmed NTM patients from the collaborating network for prospective biospecimen collection.
5. Methods and Procedures

   * Part 1 (Retrospective Survey): Data on demographics, clinical symptoms, imaging features (chest CT), microbiology, treatment regimens, and outcomes will be extracted from electronic health records. Statistical analyses will include descriptive summaries, correlation studies, and multivariable regression modeling to identify prognostic factors.
   * Part 2 (Prospective Study): Peripheral blood and bronchoalveolar lavage fluid (BALF) will be collected. Analyses will include:

   Molecular Biology: Real-time quantitative PCR for cytokine expression profiling; Western blot for protein-level assessment.

   Single-Cell Sequencing: To delineate immune cell composition, transcriptional states, and cell-cell interaction networks within the pulmonary immune microenvironment.
6. Statistical Analysis For Part 1, appropriate statistical tests (e.g., Chi-square, t-test, ANOVA, Kaplan-Meier survival analysis, Cox regression) will be applied based on data types and distribution. For Part 2, bioinformatics pipelines specific for single-cell RNA sequencing data will be employed for clustering, differential expression, and pathway analysis. A p-value <0.05 will be considered statistically significant.
7. Ethics and Data Management The study protocol will be submitted for approval to The Eighth Affiliated Hospital of Sun Yat-Sen University Ethics Committee of all participating centers prior to initiation. Patient informed consent will be obtained for the prospective Part 2. All data will be de-identified, coded, and stored on secure, password-protected servers in compliance with data protection regulations.
8. Significance This study is expected to generate a comprehensive clinical profile of NTM lung disease in South China and provide novel insights into its pathogenesis at the immune-microenvironment level. The findings may contribute to more accurate diagnostic criteria, prognostic models, and inform the future development of targeted therapeutic strategies for this refractory infection.

ELIGIBILITY:
Inclusion Criteria:1. (Both Cohorts):

* Patients diagnosed with nontuberculous mycobacterial according to standard guidelines.
* Aged 18 years or older.
* Available medical records covering the period from 2015 to 2025 (for the retrospective cohort).

  2. (Prospective Sub-cohort Additional):
* Willing and able to provide written informed consent for biospecimen collection.
* Clinically stable and suitable for undergoing research bronchoalveolar lavage (BAL) procedure, as judged by the investigator.

Exclusion Criteria: 1. (Both Cohorts):

* Active tuberculosis or other dominant pulmonary infections.
* Incomplete medical records that preclude adequate data extraction (for retrospective analysis).

  2. (Prospective Sub-cohort Additional):
* Contraindications to bronchoscopy or BAL procedure.
* Pregnancy or lactation.
* Any condition that, in the opinion of the investigator, would compromise patient safety or data integrity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population comprises patients diagnosed with nontuberculous mycobacterial infection in South China. It includes two nested cohorts: (1) a large multicenter retrospective cohort of approximately 1,500 patients identified from hospital records between 2015 and 2025, from whom clinical and epidemiological data will be extracted; and (2) a prospective sub-cohort of about 106 patients consecutively enrolled from the aforementioned group, who will provide additional biospecimens (peripheral blood and bronchoalveolar lavage fluid) for mechanistic laboratory investigations.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Phenotype Distribution | At time of diagnosis (assessed retrospectively from medical records between January 2015 and May 2025)
  Proportion of patients with different clinical-radiological phenotypes of NTM-LD (nodular-bronchiectatic, fibrocavitary, hypersensitivity-like, and mixed patterns) based on chest CT imaging and clinical presentation.
Treatment Response Categories | 12 months post-diagnosis (assessed retrospectively from medical records between January 2015 and May 2025)
  Distribution of treatment outcomes including: (1) microbiological conversion (negative cultures for ≥12 months), (2) treatment failure (persistent positive cultures despite appropriate therapy), (3) treatment intolerance requiring discontinuation, and (4) spontaneous improvement without treatment.

SECONDARY OUTCOMES:
Spectrum of NTM Species | Species distribution will be assessed at baseline, defined as the date of the first positive NTM culture from a respiratory specimen. Retrospective data collection will cover the period from January 2015 to May 2025.
  The spectrum and relative frequency of nontuberculous mycobacteria (NTM) species isolated from respiratory specimens (including sputum and bronchoalveolar lavage fluid) will be determined through retrospective analysis of positive culture and species identification results from the hospital's microbiology laboratory database. All patients with confirmed NTM pulmonary disease will be included in this analysis.
Clinical Prognostic Factors | Assessed at baseline (within 7 days of enrollment).
  Specific clinical variables assessed for their association with treatment outcome. These include: presence of cavitation on baseline chest CT, body mass index (BMI) < 18.5 kg/m² at diagnosis, CCI, NLR, NMLR, and a history of previous NTM treatment failure.
Immunological Prognostic Factors | Serum sample collected at baseline (within 7 days of enrollment) for antibody testing.
  Specific immunological variables assessed for their association with treatment outcome. This primarily refers to the presence and titer of neutralizing anti-interferon-gamma autoantibodies (nIFN-γ-autoAbs) in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Jianquan Zhang, Study Chair — The Eighth Affiliated Hospital of Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared?
  • De-identified individual participant data that underlie the results reported in the primary publication (including baseline characteristics, primary and secondary outcome measures).
  What other documents will be available?
  • Study protocol, statistical analysis plan, and informed consent form (if applicable).
  When will data be available (start and end dates)? • Beginning 1year after the publication of the primary results and ending 5 years thereafter.
  With whom? • Researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal.
  For what types of analyses?
  • For individual participant data meta-analysis or other secondary analyses approved by the proposal assessment committee.
  By what mechanism will data be made available?
  • Proposals should be directed to [principal investigator's email address, jqzhang2002@126.com]. To gain access, requestors will need to sign a data access agreement. Data will be shared v
Supporting Information: Study Protocol
Time Frame: Beginning 1year after the publication of the primary results and ending 5 years thereafter.
Access Criteria: 1. Access will be granted to external researchers (including individuals affiliated with academic institutions, healthcare organizations, or non-commercial research entities) who provide a methodologically sound research proposal that has received ethical approval (if applicable) from an institutional review board. The proposal must align with the original study's ethical framework and informed consent provisions. Proposals for commercial purposes will not be considered.
  2. Requestors may access the following de-identified datasets and documents:
  1. Individual Participant Data: Key de-identified variables including demographics (age, gender), clinical characteristics (symptoms, imaging phenotypes, NTM species), laboratory results, and primary/secondary outcome measures.
  2. Supporting Documents: The final approved study protocol, the statistical analysis plan, the informed consent form template, and the data dictionary defining all variables.
URL: https://www.icmje.org/recommendations/browse/publishing-and-editorial-issues/clinical-trial-registration.html